CLINICAL TRIAL: NCT03079232
Title: In Vivo Imaging Innovation : Optical Coherence Microscopy in Dermato-oncology
Brief Title: First Optical Coherence Microscopy in Dermato-oncology
Acronym: GALAXY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: DAMAE Médical (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1608015; 2016-A00319-42 (Other: ANSM)
Record Dates: First submitted 2016-03-16; First posted 2017-03-14 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Skin Cancer
Keywords: Optical biopsy; Skin cancer; Diagnostic performance
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Intervention Model Description: One group of patients One group of non skin cancer patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OCTAV Patient (Experimental): The patients who will have a biopsy of skin suspected to be a melanoma, basal cell carcinoma or squamous cell carcinoma will have a skin imaging with a new Microscopy Optical Coherence (OCTAV)
  Interventions: Device: OCTAV Patient
- OCTAV Control group (Experimental): Control group (patients without skin cancer) will have a skin imaging with a new Microscopy Optical Coherence (OCTAV)
  Interventions: Device: OCTAV Control group

INTERVENTIONS:
Device: OCTAV Patient — In vivo skin imaging performed by placing the tip of the OCTAV device directly in slight contact with the skin of the patient.
  Other Names: OCTAV, DAMAE Medical, Paris, France
  Arms: OCTAV Patient
Device: OCTAV Control group — In vivo skin imaging performed by placing the tip of the OCTAV device directly in slight contact with the skin of the patient.
  Other Names: OCTAV, DAMAE Medical, Paris, France
  Arms: OCTAV Control group

SUMMARY:
OCTAV is a medical device class I, not CE marked, based on a new technique for high-resolution imager (cell) internal microstructures of all types of biological tissues in vivo or ex vivo, to a depth of penetration 800 .mu.m. It allows to explore the epidermis, the dermo-epidermal junction and middle dermis in a totally non-invasive (direct contact with the tissue without sampling).

DETAILED DESCRIPTION:
At the coming of the patient in Dermatology for resection / biopsy of the tumor (usual practice), for the study, an image of the tumor will be performed with the OCTAV device (about 5 minutes) for the study. Then, according to usual practice, resection / biopsy will be performed.

This study aims to validate the clinical relevance of this device to characterize the 3 main skin cancers and to obtain the necessary data for the implementation of future clinical trials.

ELIGIBILITY:
FOR PATIENT

Inclusion Criteria:

* Patient with a cutaneous lesion suspicious for melanoma, basal cell carcinoma, squamous cell carcinoma, requiring a surgical excision
* Consent form signed
* Major patient

Exclusion Criteria:

* Allergy or intolerance to immersion oil (used for microscopy)
* If female, pregnant or breast-feeding
* Patient unable to stand still for 60 seconds
* Skin lesions located near patient eyes (<3 cm)

FOR CONTROL GROUP

Inclusion Criteria:

* Aged between 18 to 40 years
* Consent form signed
* Patient of the dermatology department with non-pathological forearm skin

Exclusion Criteria:

* Allergy or intolerance to immersion oil (used for microscopy)
* If female, pregnant or breast-feeding
* Patient unable to stand still for 60 seconds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity | Day 1
  Sensitivity measures the proportion of positive skin cancers (according to the OCTAV device) that are correctly identified as such (according to gold standard : histology)
Specificity | Day 1
  Specificity measures the proportion of negative skin cancers (according to the OCTAV device) that are correctly identified as such (according to gold standard : histology)

SECONDARY OUTCOMES:
Measure of the thickness of the different skin layers (mm) | Day 1
  Only for the non skin cancer group. Theses measures will identify the different skin layers (Epidermis, Dermis, Subcutaneous tissue, Cross-section)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc PERROT, MD, Principal Investigator — CHU SAINT-ETIENNE; Cécile DUPONT, PhD, Study Chair — Damae Medical
Locations (1):
- Chu de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No